CLINICAL TRIAL: NCT03550105
Title: Effects of Simulated Passive Jogging Device on Glucose Homeostasis, Muscle Strength and Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sackner Wellness Products LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GJHP03122018
Record Dates: First submitted 2018-05-01; First posted 2018-06-08 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Glucose Metabolism Disorders; Physical Activity
Keywords: Glucose; Diabetes; Physical Activity; Passive Exercise; Blood Pressure; Muscle Strength; Muscle Endurance; Hypertension; Physical Inactivity
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Motor Activity; Hypertension; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A) Study Subjects with Baseline Glucose of > 150mg/dl, will have Gentle Jogger Only for 7 days B) Study Subjects with Baseline Glucose of < 150 mg/dl will have basal oral glucose tolerance test (OGTT) and repeat OGTT after 7 days of Gentle Jogger
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GJ-Only (Experimental): Study Subjects with Baseline Glucose of > 150mg/dl, will have Gentle Jogger Only for 7 days
  Interventions: Device: Gentle Jogger
- GJ-OGTT (Experimental): Study Subjects with Baseline Glucose of < 150mg/dl, will have Oral Glucose Tolerance Test (OGTT) at baseline and after 7 days of Gentle Jogger
  Interventions: Device: Gentle Jogger

INTERVENTIONS:
Device: Gentle Jogger — Gentle Jogger is a passive simulated jogging device to be used 3 times per day for at least 30 mins for 7 days in this study

SUMMARY:
Physical Inactivity and excessive sedentary behavior are risk factors for diabetes and cardiovascular disease. Movement is important for overall health. This study will assess the validity and usefulness of low risk, non-invasive wellness device, the Gentle Jogger® (GJ) that passively simulates the physical activities of jogging. The study will evaluate whether or not use of GJ modifies glycemic control and muscle strength in subjects who are known to be diabetic and those who are not. The study volunteers are subjects between the ages of 25-80yr.

DETAILED DESCRIPTION:
Excessive sedentary behavior and physical inactivity are independent risk factors for; obesity, metabolic syndrome, heart disease, Type 2 Diabetes Mellitus (T2DM), and hypertension. In adults with T2DMT interrupting prolonged sitting improves glycemic control. Increasing physical activity even briefly (3-15 min) is effective in reducing postprandial hyperglycemia and improving glycemic control. To address the excessive sedentary behavior Sackner Wellness Products has patented a non-invasive method for inducing passive movement while in seated or supine posture the Gentle Jogger® (GJ)which simulates the activities of jogging. Passive simulation of jogging introduces pulses into the circulation as the foot strikes the device. These pulsations have been shown to elicit production of beneficial mediators which are important to cardiovascular health. The study will recruit two groups of subjects ages 25-80. One group (n=45) of either sex who are not known to be diabetics and have a normal fasting glucose. Another group (n=45) who are known to be diabetics (Type 1 or Type 2) previously diagnosed by their physician and currently on insulin and or oral medications. Exclusion criteria are those younger than 25yrs and greater than 80yrs, and inability to provide informed consent. The study will last 14 days total and will consist of 5 study visit days. Volunteers will be paid for their participation in the study.

On day 1 participants will have a continuous interstitial glucose sensor ( Freestyle Libre Pro), and an activity monitor placed. The participants will have their blood pressure measured and muscle strength and endurance measured using a dynamometer which measures grip force. Based on the average glucose obtained on day 1-2 of the study, subjects will be assigned to two groups. A) GJ-Only (subjects with baseline average glucose of > 150mg/dl or B) GJ with Oral Glucose Tolerance Testing(GJ-OGTT) (subjects with baseline average glucose of < 150mg/dl).

On day 3 those enrolled in GJ-OGTT groups will have a basal oral glucose tolerance test and grip force and blood pressure will be measure before and after the OGTT. Those enrolled in GJ -Only group will only have grip force and blood pressure measured. Day 4 of the study all subjects will be instructed on the use of GJ device and will be asked to use the device 3 times per day for 30 min, from day 4 till day 11. On day 11 those enrolled in GJ-OGTT groups will have a repeat oral glucose tolerance test , grip force and blood pressure will be measure before and after the OGTT. Those enrolled in GJ -Only group will only have grip force and blood pressure measured. On day 14 all subjects will have grip force and blood pressure measured and a brief debriefing about their experience with GJ.

The total days enrolled in the study are14 days.

The Gentle Jogger's intended use as a wellness device in which , 1) GJogger are part of a healthy lifestyle, which may help to reduce the risk of certain chronic diseases or conditions such as heart disease, high blood pressure, and type 2 diabetes and, 2) may help living well with certain chronic diseases or conditions such as s heart disease, high blood pressure, and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers able to consent ages 25-80yrs
* Known Diabetics (Type 1 or Type 2)- Previously diagnosed by their physician on either Insulin and or oral diabetic medications ages 25-80yrs

Exclusion Criteria:

* Younger than 25 yrs or Older than 80 yrs
* Unable to provide consent

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 8 days
  For GJ-OGTT Group: Blunting of the peak and decrease of the area under the curve of the Oral Glucose Tolerance after 7 days of Gentle Jogger For GJ-Only Blunting or decreased of basal glucose levels ( 3 days prior to GJ) compared to glucose levels after 7 days of GJ

SECONDARY OUTCOMES:
Variability of Glycemic Control - (24 hrs Standard Deviation of Glycemia) | 8 Days
  Comparison of 24 hrs of Glycemic variability at 3 time periods a)24 hrs before GJ b) the last 24 hrs of GJ and c) Last 24 hrs of study ( day 13-14)
Muscle Strength | 8 days
  For GJ-OGTT Group: improved grip force after 7 days of GJ Compared to prior to GJ For GJ-Only improved grip force after 7 days of GJ Compared to prior to GJ
Muscle Endurance | 8 days
  For GJ-OGTT Group: improved grip endurance after 7 days of GJ Compared to prior to GJ For GJ-Only improved grip force and endurance after 7 days of GJ Compared to prior to GJ
Carry Over Effect of Muscle Strength | 14 days
  For BOTH Groups: Comparison of grip force between last day of GJ and day 14 ( 3 days after completion of GJ)
Carry Over Effect of Muscle Endurance | 14 days
  For BOTH Groups: Comparison of muscle strength between last day of GJ and day 14 ( 3 days after completion of GJ)

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams JA, Lopez JR, Nadkarni V, Zolkipli-Cunningham Z, Ischiropoulos H, Sackner MA. The effects of a motorized passive simulated jogging device on descent of the arterial pulse waveform dicrotic notch: A single arm placebo-controlled cross-over trial. Physiol Rep. 2022 Aug;10(15):e15418. doi: 10.14814/phy2.15418. PMID 35924333
- [Derived] Adams JA, Lopez JR, Banderas V, Sackner MA. The Effects of Passive Simulated Jogging on Parameters of Explosive Handgrip in Nondiabetics and Type 2 Diabetics: A Single Arm Study. Biomed Res Int. 2022 Feb 11;2022:6450844. doi: 10.1155/2022/6450844. eCollection 2022. PMID 35187168
- [Derived] Adams JA, Lopez JR, Banderas V, Sackner MA. A single arm trial using passive simulated jogging for blunting acute hyperglycemia. Sci Rep. 2021 Mar 19;11(1):6437. doi: 10.1038/s41598-021-85579-7. PMID 33742027
- [Derived] Adams JA, Banderas V, Lopez JR, Sackner MA. Portable Gentle Jogger Improves Glycemic Indices in Type 2 Diabetic and Healthy Subjects Living at Home: A Pilot Study. J Diabetes Res. 2020 Jan 21;2020:8317973. doi: 10.1155/2020/8317973. eCollection 2020. PMID 32215273